CLINICAL TRIAL: NCT05958069
Title: The Efficacy and Safety of Minocycline in the Treatment of Drug-resistant Epilepsy in NORSE Patients: an Open-label, One-arm Clinical Study
Brief Title: The Efficacy and Safety of Minocycline in the Treatment of Drug-resistant Epilepsy in NORSE Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Li Hui, Director, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJLL-KY-20232108
Record Dates: First submitted 2023-04-13; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Epileptic Seizures Related to Drugs
MeSH Terms: interventions — Minocycline; Anticonvulsants

STUDY DESIGN:
Intervention Model Description: Treatment with minocycline combined with antiepileptic drugs: After enrollment, 100mg/day (50mg specification) of minocycline hydrochloride was administered for 12 consecutive weeks;
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- minocycline (Experimental): Treatment with minocycline combined with antiepileptic drugs: After enrollment, 100mg/day (50mg specification) of minocycline hydrochloride was administered for 12 consecutive weeks;
  Interventions: Drug: minocycline

INTERVENTIONS:
Drug: minocycline — Treatment with minocycline combined with antiepileptic drugs: After enrollment, 100mg/day (50mg specification) of minocycline hydrochloride was administered for 12 consecutive weeks;
  Other Names: antiepileptic drugs

SUMMARY:
Exploring the efficacy and safety of oral minocycline combined with antiepileptic drugs in the treatment of drug-resistant epilepsy in NORSE patients, obtaining preliminary research data, and providing evidence and data support for the next large-scale randomized controlled clinical study.

DETAILED DESCRIPTION:
New-onset refractory status epilepticus (NORSE) is a rare but special clinical manifestation with a high mortality rate. Most cases evolve into Super refractory status epilepticus (SRSE), with poor treatment efficacy, short-term mortality rate of 12-27%, and high long-term disability rate. Most survivors eventually develop into Drug resistant epilepsy (DRE) and experience cognitive impairment. Frequent seizures seriously affect patients' daily life and work, Controlling the frequency of seizures is particularly important. At present, the pathogenesis of this disease is still unclear, and the treatment plan is still controversial. In recent years, research has found that inflammatory and immune responses in the body may be involved in the pathogenic process. In response to the current research on the inflammatory immune mechanism and epilepsy, the use of anti-inflammatory drugs and immune modulators may be a new treatment direction.

Minocycline is a semi synthetic tetracycline broad-spectrum antibiotic with good blood-brain barrier penetration. Since the end of the 19th century, the efficacy of minocycline has been reported in many models of nervous system disease, including hemorrhagic and ischemic stroke, multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease, etc. Because of its ability to cross the blood-brain barrier, its detoxification effect on activated microglia and its proven human safety record, it seems to be a promising candidate drug for epilepsy treatment.

In summary, minocycline has good blood-brain barrier permeability, as well as anti-inflammatory, immunomodulatory, and potential anti epileptic effects, with good safety. Therefore, this study intends to carry out a randomized controlled, open label, evaluator blind proof of concept study to explore the efficacy and safety of minocycline in the treatment of drug-resistant epilepsy in patients with NORSE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 8 years old;
2. It meets the NORSE diagnostic criteria: (1) newly emerging intractable status epilepticus, (2) no previous epilepsy or other related nervous system disease, (3) no clear acute structural, toxic and metabolic factors leading to intractable status epilepticus;
3. NORSE medical history ≥ 6 months, with a frequency of ≥ 4 episodes per month;
4. Take two or more antiepileptic drugs;
5. The patient and their family members are aware of this study and sign an informed consent form.

Exclusion Criteria:

1. Patients who are allergic to any component of tetracycline or product formulation;
2. Persistent state of epilepsy;
3. Adjustment of antiepileptic drugs during the trial period;
4. Immunotherapy, ketogenic diet and other added treatments were not stable or other treatments were started during the trial;
5. Epilepsy surgery;
6. In the treatment of vagus nerve stimulation and transcranial magnetic stimulation;
7. Patients with severe infection, cerebrovascular disease, malignant tumor and other nervous system disease, and patients with severe dysfunction of heart, liver, kidney and other organs;
8. Non epileptic seizures such as syncope and hysteria;
9. Participating in clinical trials of other drugs;
10. Women during lactation or pregnancy;
11. Incomplete clinical data;
12. The patient or family member withdraws the informed consent form.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in seizure frequency | 24 months
  Main efficacy endpoint: Changes in seizure frequency from baseline in patients who added minocycline during the 12 week treatment period. Epileptic seizures include countable focal motor seizures with unconscious disorders, focal seizures with conscious disorders, focal seizures evolving into bilateral motor seizures, and systemic seizures (tonic-clonic, tonic-clonic, or atonic);
Incidence of adverse events (Main safety indicators) | 24 months
  such as dizziness, rash, and gastrointestinal reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Wen jiang, Study Chair — The First Affiliated Hospital of Air Force Military Medical University; Lei Ma, Principal Investigator — The First Affiliated Hospital of Air Force Military Medical University; yuanyuan Wang, Principal Investigator — XijingHospital; mengmeng Hu, Principal Investigator — XijingHospital
Locations (1):
- XijingHospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Feng L, Li H, Ma L, Hu M, Hui B, Sun Z, Wang X, Wang Y, Jiang W. Minocycline in chronic management of febrile infection-related epilepsy syndrome (FIRES): a case series and literature review of treatment strategies. Acta Epileptol. 2025 Jun 6;7(1):35. doi: 10.1186/s42494-025-00224-4. PMID 40481521